CLINICAL TRIAL: NCT03131765
Title: Phase 1, Open Label, Dose Escalation and Cohort Expansion Study of YS-ON-001 in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation and Cohort Expansion Study of YS-ON-001 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YS-RVON-001
Record Dates: First submitted 2017-03-07; First posted 2017-04-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: YS-ON-001 is a single agent used for this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YS-ON-001 (Experimental): Phase 1- Dose escalation based on YS-ON-001 safety and tolerability obtained from three subjects enrolled in a cohort (first cycle of treatment), enrollment at the next dose level or additional subjects into the ongoing cohort will occur.
  Phase 1b- recommended dose determined in Phase 1. Enrollment of two expansion cohorts will be restricted to the tumour types, breast cancer and liver cancer
  Interventions: Biological: YS-0N-001

INTERVENTIONS:
Biological: YS-0N-001 — Cancer vaccine
  Other Names: Polyinosinic-polycytidylic acid/inactivated rabies virus

SUMMARY:
Phase 1 study evaluating the safety and tolerability of YS-ON-001 in patients with advanced solid tumors who have limited available treatment options, and exploratory evaluation of the pharmacological effect and efficacy of YS-ON-001. The study will be conducted in two parts: dose escalation and cohort expansion

DETAILED DESCRIPTION:
This is an open-label, Phase 1 study of YS-ON-001 vaccine administered intramuscularly (IM) as a single agent to patients with advanced solid tumors. Patients are eligible if they are refractory, resistant or intolerant to prior therapies.The study will assess YS-ON-001 administered as a single agent, three times per week for 21-days with 1 week wash out period (28 days as 1 cycle) for 12 cycles in a continuous regimen. A dose escalation design will be applied in cohorts of 3-6 patients in Part I of the study.

The starting dose will be 2ml (3 times/ week). Once the recommended phase II dose (RP2D) is established, the cohort will be expanded with at least 10 additional patients to further characterize the safety and tolerability at RP2D with specific tumour types, Breast cancer and Liver Cancer

Treatment with YS-ON-001 may be continued for up to 12 cycles or until disease progression or if patient is withdrawn or unacceptable toxicity occurs. Patients who complete 12 cycles of treatment will be considered to have completed the trial. Patients who continue to benefit from treatment after 12 cycles may have the option to continue treatment upon agreement between the investigator and sponsor, and pending study drug availability.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 3 months
* Patient with histologically or cytologically proven advanced (unresectable) or metastatic solid tumor who have failed standard therapies or are intolerant to standard therapies.Part 1: Any advanced or metastatic solid tumor patient Part 2: Selected tumor types including cytological or histologically diagnosed breast cancer and liver cancer
* Patients with adequate bone marrow function, with absolute neutrophil count (ANC) >1,500/mm3, platelet count >100,000/mm3, and hemoglobin > 10 g/mm3
* Patients with adequate kidney function, with serum creatinine ≤1.5 X upper limit of normal (ULN)
* Patients with adequate liver function, with aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x ULN, total bilirubin ≤1.5x ULN ; For patients with liver metastasis, AST, ALT ≤5x ULN, Total bilirubin ≤1.5x ULN
* Patients with adequate coagulation function, with activated partial thromboplastin time (aPTT) ≤1.5x ULN
* Female patients, if of childbearing potential, must have a negative serum pregnancy test within 72 hours prior to the date of the first dose of study medication.
* Female patients of childbearing potential and male patients must agree to use adequate methods of contraception with their partner starting with the screening visit up to 4 weeks after the last dose of study therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.

Exclusion Criteria:

* Known uncontrolled seizures, central nervous system disorders, or loss of cognitive ability due to mental illness
* Pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study.
* Patient is currently receiving or has received systemic corticosteroids within 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. The following use of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airway diseases), eye drops or local injections (e.g., intra-articular).
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Known serious, uncontrolled medical conditions that in the opinion of the investigator, will render it unsafe for the patient to receive the study therapy
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Patient has not recovered (i.e., to ≤ Grade 1 or to baseline) from radiation- and chemotherapy-induced adverse events (AEs) or administration of colony-stimulating factors (including granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF) or recombinant erythropoietin) within 3 weeks prior to the first dose of study drug.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational drug within 4 weeks prior to the first dose of study drug.
* Received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 21 days, or less than 5 times the half-life of the most recent therapy prior to study Day 1, whichever is shorter. Note: palliative radiation therapy to a small field ≥ 1 week prior to Day 1 of study treatment will be allowed.
* Patient has not recovered adequately (≤ Grade 1) from AEs and/or complications from any major surgery prior to starting therapy. Patient has received a vaccine within 7 days of planned start of study therapy.
* Known hypersensitivity to YS-ON-001 components or excipients
* Known unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction that occurred within a year, severe arrhythmia that required drug treatment, liver disease, kidney disease and metabolic diseases)
* Known history of splenectomy
* Known history of chronic alcohol or drug abuse within 6 months
* PI assessment of subject's lack of willingness to participate and comply with all requirements of the protocol
* Any other finding which, in the opinion of the PI would significantly increase the risk of having an adverse outcome from participating in this protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Safety of YS-ON-001 by monitoring any adverse events (AE) and serious adverse events (SAE) | through study completion, an average of 1 year
  To assess the safety of YS-ON-001 in patients with advanced (metastatic and/or unresectable) solid tumors based on the identification of any adverse events through study completion
Tolerability of YS-ON-001 by recording AE /SAE, clinically significant changes in lab parameters and performance status (ECOG) | 6 months
  To assess the tolerability of YS-ON-001 in patients with advanced (metastatic and/or unresectable) solid tumors for recommended phase II dose (RP2D)
Dose-limiting toxicities (DLT) | For 4 weeks for DLTs
  Number of Participants with a Dose Limiting Toxicity (DLT)

SECONDARY OUTCOMES:
Antitumor Activity of YS-ON-001 by imaging measurement and assessing using RECIST Version 1.1 | At 2 months, 4 months., 6months, 9 months and 1 year
  Assessment of antitumor activity of YS-ON-001 in advanced solid tumors based on the change of response rate on RECIST v1.1 at 2 months, 4 months., 6months, 9 months and 1 year
Immunogenicity of YS-ON-001 evaluated by measuring serum titre level antibody against YS-ON-001 | At 3 months, 6 months, 9 months and 1 year
  To observe immune response in patients administered with YS-ON-001

CONTACTS AND LOCATIONS:
Overall Officials: Lee Soo Chin, Principal Investigator — National University of Singapore
Locations (1):
- National University Cancer Institute Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No